CLINICAL TRIAL: NCT07100093
Title: Prospective, Multicenter Study on the Association Between Serum Ustekinumab Levels and Clinical, Biological and Endoscopic Remission in Patients With Crohn's Disease.
Acronym: USTECRO
Status: Completed | Type: Observational
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, María Dolores Martín Arranz, PhD, Principal Investigator, Hospital Universitario La Paz
Other Study IDs: PI-4732
Record Dates: First submitted 2025-07-30; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Ustekinumab Serum Levels in Patients With Crohn´s Disease
Keywords: Ustekinumab; Serum levels; Crohn´s disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Induction: Patients with an established diagnosis of Crohn's disease according to the usual criteria (clinical, analytical, endoscopic, radiological and/or histological) with inflammatory activity, who initiate treatment with ustekinumab for induction of remission. Activity will be considered the presence of clinical activity (Harvey-Bradshaw index ≥5) and/or elevation of fecal calprotectin (≥ 250µg/g; ≥100 in case of interventional CD) and/or presence of endoscopic activity (SES-CD ≥3).
  Interventions: Procedure: Drug serum levels
- Maintenance: Patients with an established diagnosis of Crohn's disease according to usual criteria (clinical, analytical, endoscopic, radiological and/or histological) on maintenance treatment with ustekinumab stably for a minimum of 6 months.
  Interventions: Procedure: Drug serum levels

INTERVENTIONS:
Procedure: Drug serum levels — Ustekinumab trough levels (prior to administration of the next dose of the drug) will be determined by enzyme-linked immunoadsorption assay (ELISA) methodology.

SUMMARY:
A prospective, non-commercial, multicenter study will be conducted in a cohort of patients initiating induction therapy and a cohort of patients with stable treatment with ustekinumab.

DETAILED DESCRIPTION:
The present study aims to evaluate the association between serum levels (trough) of Ustekinumab and clinical, biological, endoscopic and radiological response/remission in patients with Crohn's disease, in order to determine threshold levels at induction and maintenance that may be predictors of efficacy.

Working hypothesis: Serum Ustekinumab levels in Crohn's disease patients are correlated with clinical, biochemical and endoscopic/radiological response/remission.

Patients with an established diagnosis of Crohn's disease by usual criteria (clinical, analytical, endoscopic, radiological and/or histological) who initiate treatment with Ustekinumab (induction cohort) or who are on maintenance treatment with Ustekinumab (maintenance cohort) in a stable dosis (a minimum of 6 months) will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an established diagnosis of CD according to standard criteria (clinical, analytical, endoscopic, radiological, and/or histological) with inflammatory activity, who begin treatment with ustekinumab for remission induction. Activity will be considered to be the presence of clinical activity (Harvey-Bradshaw index ≥5) and/or elevated fecal calprotectin (≥ 250μg/g; ≥100 in cases of surgically treated CD) and/or the presence of endoscopic activity (SES-CD ≥3).
* Patients with a confirmed diagnosis of CD according to standard criteria (clinical, analytical, endoscopic, radiological, and/or histological) undergoing stable maintenance treatment with ustekinumab for at least 6 months.

Exclusion Criteria:

* Patients in whom ustekinumab is indicated for the prevention of post-surgical recurrence.
* Patients in whom ustekinumab is indicated for the control of perianal disease.
* Patients in whom ustekinumab is indicated for the control of extraintestinal manifestations.
* Pregnant women.
* Patients who are unable to understand the nature of the study, the procedures to be followed, or who are not able to sign an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an established diagnosis of CD based on standard criteria (clinical, laboratory, endoscopic, radiological, and/or histological) who are starting treatment with ustekinumab (induction cohort) or who are undergoing maintenance treatment with ustekinumab (maintenance cohort) on a stable basis (minimum of 6 months) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
biological remission | week 8 and week 16
  association between serum levels of ustekinumab and biological remission in induction

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No